CLINICAL TRIAL: NCT03876613
Title: Comparison of Different Music Types in Reducing Dental Anxiety in Young People Undergoing Third Molar Tooth Surgery - A Randomized Controlled Study
Brief Title: Different Music Types in Reducing Dental Anxiety in Young People
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Erzincan University (Other)
Responsible Party: Principal Investigator, ILKE KUPELI, assist. prof., Erzincan University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: EBYU
Record Dates: First submitted 2019-03-08; First posted 2019-03-15 (Actual); Last update posted 2019-07-16 (Actual); Status verified 2019-07

CONDITIONS: Dental Anxiety

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Turkish music group (Active Comparator): Rast makam
  Interventions: Behavioral: Different music types
- classical western music (Active Comparator): Vivaldi
  Interventions: Behavioral: Different music types
- soft rock music (Active Comparator): Elvis presley
  Interventions: Behavioral: Different music types
- control group (Placebo Comparator): No music
  Interventions: Behavioral: Different music types

INTERVENTIONS:
Behavioral: Different music types — the type of music that reduces anxiety best and most effectively.

SUMMARY:
Anxiety is an important issue in dental care for adults, children and adolescents. Dental anxiety affects 10-20% of adults and 43% of children and adolescents. Dental anxiety often leads to avoiding dental treatment; this can cause serious deterioration of oral and dental health. Such deterioration can significantly increase dental care costs. Therefore, reducing anxiety is important both in terms of patient, physician and cost. Music intervention is a psychological therapy that has many advantages when used in outpatient treatment, including cost-effectiveness, lack of negative physical effects, rapid effect, lack of safety in terms of non-use and lack of concern for recovery. Some types of studies suggested but not tested against each other include classical music, soft rock, calming music, pop, easy listening music, and music of choice.

With the contradictory results of various studies, the fact that the distraction of music and its distraction on the reduction of tooth anxiety is not common shows that a more structured study is needed. The lack of precise data on the effects of different music types on anxiety has led to this study.

ELIGIBILITY:
Inclusion Criteria:

* 3. Molar tooth extraction,
* 18-30 years old,
* Symptomatic

Exclusion Criteria:

* Who does not agree to participate in the study,
* Under 18 years, over 30 years,
* patients with impaired hearing (ie, not suitable for musical intervention),
* arrhythmia
* patients with physical condition III or higher (American Society of Anesthesiologists)

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-07-15 (Estimated); Primary Completion 2019-12-15 (Estimated); Study Completion 2020-01-15 (Estimated)

PRIMARY OUTCOMES:
Number of the patients with anxiety | six month
  the type of music that reduces anxiety best and most effectively.

CONTACTS AND LOCATIONS:
Overall Officials: ilke kupeli, Principal Investigator — Erzincan University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Almoznino G, Zini A, Sharav Y, Shahar A, Zlutzky H, Haviv Y, Lvovsky A, Aframian DJ. Sleep quality in patients with dental anxiety. J Psychiatr Res. 2015 Feb;61:214-22. doi: 10.1016/j.jpsychires.2014.11.015. Epub 2014 Dec 9. PMID 25529787
- [Result] Gordon D, Heimberg RG, Tellez M, Ismail AI. A critical review of approaches to the treatment of dental anxiety in adults. J Anxiety Disord. 2013 May;27(4):365-78. doi: 10.1016/j.janxdis.2013.04.002. Epub 2013 Apr 13. PMID 23746494
- [Result] Shim YS, Kim AH, Jeon EY, An SY. Dental fear & anxiety and dental pain in children and adolescents; a systemic review. J Dent Anesth Pain Med. 2015 Jun;15(2):53-61. doi: 10.17245/jdapm.2015.15.2.53. Epub 2015 Jun 30. PMID 28879259